CLINICAL TRIAL: NCT05778396
Title: Feasibility of Blinding Spinal Manual Therapy Interventions for a Trial Assessing Management of Primary Care Patients With Back Pain: the SALuBRITY Blinding Feasibility Randomised Controlled Trial
Brief Title: Feasibility of Spinal Manual Therapy Interventions for a Future Clinical Study of Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balgrist University Hospital (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Principal Investigator, Cesar A Hincapié, DC PhD, Senior Scientist and Head of Musculoskeletal Epidemiology Research, Balgrist University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: SALuBRITY Blinding
Record Dates: First submitted 2023-02-27; First posted 2023-03-21 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-06

CONDITIONS: Back Pain; Back Pain With Radiation; Back Pain, Low
Keywords: Methods; Manual therapy; Randomized trial; Back pain; Blinding assessment
MeSH Terms: conditions — Back Pain; Low Back Pain

STUDY DESIGN:
Intervention Model Description: Two-parallel-group, single-centre, sham-controlled, methodological blinding feasibility randomised trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, managing clinicians, outcome assessors, data analysts, and investigators will be blinded to intervention assigned. Only treating clinicians will not be blinded to the interventions but will be trained and asked not to disclose the intervention, nature of the interventions, nor trial objectives to trial participants or other members of the trial team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active spinal manual therapy protocol (Active Comparator): (1) Side-lying lumbar spine manipulation, (2) prone lumbar spine mobilization, and (3) prone thoracic spine manipulation.
  Interventions: Procedure: Active spinal manual therapy protocol
- Control spinal manual therapy protocol (Sham Comparator): (1) Control side-lying lumbar spine manipulation, (2) control prone lumbar spine mobilization, and (3) control prone thoracic spine manipulation.
  Interventions: Procedure: Control spinal manual therapy protocol

INTERVENTIONS:
Procedure: Active spinal manual therapy protocol — The chiropractor will start by (1) placing one hand over L4-L5 or L5-S1 and then will apply a high-velocity, low-amplitude (HVLA) thrust with a therapeutic line of drive. Side-lying lumbar manipulation will be performed bilaterally, with the treating clinician choosing any suitable technique and with or without occurrence of the characteristic audible joint cavitation associated with spine manipulation. The chiropractor will then perform (2) prone lumbar mobilisation by placing the contact hand and applying downward pressure over L4-L5 or L5-S1 with the other hand guiding a manual flexion-distraction piece to apply therapeutic mobilization of the lumbar spine. The chiropractor will deliver (3) a prone thoracic manipulation by placing two hands over the transverse processes of T5-T6 or T6-T7 and applying a HVLA thrust in a posterior-to-anterior direction.
  Arms: Active spinal manual therapy protocol
Procedure: Control spinal manual therapy protocol — (1) Control side-lying lumbar manipulation will be operationalised as the application of a low-velocity broad push manoeuvre to the gluteal region following a non-therapeutic line of drive. The chiropractor will then perform (2) control prone lumbar mobilisation, consisting of a non-therapeutic manual manoeuvre involving minimal oscillations (0 to ±2°) of the flexion-distraction piece with light touch over the lumbar spine region, and (3) control prone thoracic mobilisation consisting of two-handed left and right scapula pushes with a nontherapeutic line of drive.
  Arms: Control spinal manual therapy protocol

SUMMARY:
This study aims to compare two different spinal manual therapy interventions of the back to determine if they are viable and acceptable for a future study investigating the treatment of patients with back pain. The two proposed spinal manual therapy interventions are widely used in the fields of chiropractic, physical therapy, osteopathy, and manual medicine to treat back pain and improve function. This is a randomized study, meaning that participants are randomly assigned (like tossing a coin) to one of two manual spinal therapy interventions.

DETAILED DESCRIPTION:
Clinical trials of spinal manual therapy interventions for back pain and back-related leg pain face methodological challenges regarding the design of effective sham control ('control' hereafter) and blinding of the assigned interventions. Although the assessment of blinding is often neglected in the field of manual medicine, the implementation of high-quality trials of spinal manual therapy interventions warrants formal evaluation of blinding feasibility among participants and outcome assessors to advance randomized clinical trial methods and design.

The objectives of this blinding feasibility trial are:

1. To assess the feasibility of blinding participants, with or without experience of spinal manual therapy or current low back pain, randomly allocated to an active or control spinal manual therapy intervention protocol.
2. To assess the feasibility of blinding managing clinicians (non-treating clinicians or outcome assessors) within the randomised trial context.
3. To examine the impact of spinal manual therapy experience in the past 3 months (Yes vs No) and presence of low back pain during the past four weeks (average intensity ≤2 versus ≥3 out of 10) on the feasibility of participant and managing clinician blinding.
4. To explore factors contributing to participant and managing clinician perceptions about the assigned intervention (active versus control) using a qualitative thematic analysis.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* With or without experience of spinal manual therapy
* With or without experience of current low back pain

Exclusion Criteria:

* Serious spinal pathology (e.g. spinal fracture, cancer or infection)
* History of lumbar spine surgery
* Currently under care or in consultation with a specialist, chiropractor, physiotherapist, or osteopath for current back pain
* Manual medicine health care provider (i.e., chiropractor, physiotherapist, osteopath, massage therapist, manual medicine trained physician)
* Have a serious comorbidity preventing them from attending the research clinic and receiving the interventions
* Pregnant or breastfeeding status
* Involved in pending litigation related to back pain
* Already participating in another research study related to back pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2023-04-04 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2023-04-25 (Actual)

PRIMARY OUTCOMES:
Participant blinding success, as measured by the validated Bang blinding index, immediately after intervention session 1. | Immediately after intervention session 1 (study day 1)
  The blinding assessment survey item will ask: "Which treatment do you believe you received?" with five response options provided: "Strongly believe I received the genuine treatment," "Somewhat believe I received the genuine treatment," "Somewhat believe I received the control treatment," "Strongly believe I received the control treatment," and "I do not know which treatment I received." Bang BI estimates (between -1 to +1, with 0 indicating satisfactory blinding) can be interpreted as the proportion of correct guesses beyond chance within an intervention arm. For the Bang BI, a score with an absolute value of ≤0.3 (i.e., -0.3 to 0.3) will be deemed compatible with satisfactory blinding, and blinding scenarios will be discussed.
Participant blinding success, as measured by the validated Bang blinding index, immediately after intervention session 2. | Immediately after intervention session 2 (study day 2, between 48 hours and 2 weeks after study day 1)
  The blinding assessment survey item will ask: "Which treatment do you believe you received?" with five response options provided: "Strongly believe I received the genuine treatment," "Somewhat believe I received the genuine treatment," "Somewhat believe I received the control treatment," "Strongly believe I received the control treatment," and "I do not know which treatment I received." Bang BI estimates (between -1 to +1, with 0 indicating satisfactory blinding) can be interpreted as the proportion of correct guesses beyond chance within an intervention arm. For the Bang BI, a score with an absolute value of ≤0.3 (i.e., -0.3 to 0.3) will be deemed compatible with satisfactory blinding, and blinding scenarios will be discussed.

SECONDARY OUTCOMES:
Participant blinding success, as measured by the validated James blinding index, immediately after intervention session 1. | Immediately after intervention session 1 (study day 1)
  The James BI, a modification of the kappa statistic that measures disagreement beyond chance, returns a value between 0 and 1, with 1 equal to all "don't know" responses (complete blinding), 0 equal to all correct responses (complete unblinding), and 0.5 where respondents' responses appear random (50% correct, 50% incorrect).
Participant blinding success, as measured by the validated James blinding index, immediately after intervention session 2. | Immediately after intervention session 2 (study day 2, between 48 hours and 2 weeks after study day 1)
  The James BI, a modification of the kappa statistic that measures disagreement beyond chance, returns a value between 0 and 1, with 1 equal to all "don't know" responses (complete blinding), 0 equal to all correct responses (complete unblinding), and 0.5 where respondents' responses appear random (50% correct, 50% incorrect).
Outcome assessor blinding success, as measured by the validated Bang index, immediately after intervention session 1. | Immediately after intervention session 1 (study day 1)
  Bang BI estimates (between -1 to +1, with 0 indicating satisfactory blinding) can be interpreted as the proportion of correct guesses beyond chance within an intervention arm.
Outcome assessor blinding success, as measured by the validated Bang index, immediately after intervention session 2. | Immediately after intervention session 2 (study day 2, between 48 hours and 2 weeks after study day 1)
  Bang BI estimates (between -1 to +1, with 0 indicating satisfactory blinding) can be interpreted as the proportion of correct guesses beyond chance within an intervention arm.
Outcome assessor blinding success, as measured by the validated James index, immediately after intervention session 1. | Immediately after intervention session 1 (study day 1)
  The James BI measures disagreement beyond chance and returns a value between 0 and 1, with 1 equal to all "don't know" responses (complete blinding), 0 equal to all correct responses (complete unblinding), and 0.5 where respondents' responses appear random (50% correct, 50% incorrect).
Outcome assessor blinding success, as measured by the validated James index, immediately after intervention session 2. | Immediately after intervention session 2 (study day 2, between 48 hours and 2 weeks after study day 1)
  The James BI measures disagreement beyond chance and returns a value between 0 and 1, with 1 equal to all "don't know" responses (complete blinding), 0 equal to all correct responses (complete unblinding), and 0.5 where respondents' responses appear random (50% correct, 50% incorrect).

OTHER OUTCOMES:
Lumbar spine range of motion, immediately before intervention session 1. | Immediately before intervention session 1 (study day 1)
  Maximum active total flexion and extension (0 to 100+ degrees) in standing position, measured with a validated mobile phone measuring device. Higher scores represent higher flexibility.
Lumbar spine range of motion, immediately after intervention session 1. | Immediately after intervention session 1 (study day 1)
  Maximum active total flexion and extension (0 to 100+ degrees) in standing position, measured with a validated mobile phone measuring device. Higher scores represent higher flexibility.
Lumbar spine range of motion, immediately before intervention session 2. | Immediately before intervention session 2 (study day 2, between 48 hours and 2 weeks after study day 1)
  Maximum active total flexion and extension (0 to 100+ degrees) in standing position, measured with a validated mobile phone measuring device. Higher scores represent higher flexibility.
Lumbar spine range of motion, immediately after intervention session 2. | Immediately after intervention session 2 (study day 2, between 48 hours and 2 weeks after study day 1)
  Maximum active total flexion and extension (0 to 100+ degrees) in standing position, measured with a validated mobile phone measuring device. Higher scores represent higher flexibility.
Self-rated general health, immediately before intervention session 1. | Immediately before intervention session 1 (study day 1)
  Participants will answer the question "In general, would you say your health is" with five possible ordinal answers: "Excellent," "Very good," "Good," "Fair," and "Poor" (from the PROMIS tool).
Self-rated general health, immediately after intervention session 1. | Immediately after intervention session 1 (study day 1)
  Participants will answer the question "In general, would you say your health is" with five possible ordinal answers: "Excellent," "Very good," "Good," "Fair," and "Poor" (from the PROMIS tool).
Self-rated general health, immediately before intervention session 2. | Immediately after intervention session 2 (study day 2, between 48 hours and 2 weeks after study day 1)
  Participants will answer the question "In general, would you say your health is" with five possible ordinal answers: "Excellent," "Very good," "Good," "Fair," and "Poor" (from the PROMIS tool).
Self-rated general health, immediately after intervention session 2. | Immediately after intervention session 2 (study day 2, between 48 hours and 2 weeks after study day 1)
  Participants will answer the question "In general, would you say your health is" with five possible ordinal answers: "Excellent," "Very good," "Good," "Fair," and "Poor" (from the PROMIS tool).
Pain intensity, current, immediately before intervention session 1. | Immediately before intervention session 1 (study day 1)
  Participants will answer the question "What number best describes your current mid and low back pain?". Higher values represent higher levels of pain (10 = "pain as bad as you can imagine"; 0 = "no pain").
Pain intensity, current, immediately after intervention session 1. | Immediately after intervention session 1 (study day 1)
  Participants will answer the question "What number best describes your current mid and low back pain?". Higher values represent higher levels of pain (10 = "pain as bad as you can imagine"; 0 = "no pain").
Pain intensity, current, immediately before intervention session 2. | Immediately before intervention session 2 (study day 2, between 48 hours and 2 weeks after study day 1)
  Participants will answer the question "What number best describes your current mid and low back pain?". Higher values represent higher levels of pain (10 = "pain as bad as you can imagine"; 0 = "no pain").
Pain intensity, current, immediately after intervention session 2. | Immediately after intervention session 2 (study day 2, between 48 hours and 2 weeks after study day 1)
  Participants will answer the question "What number best describes your current mid and low back pain?". Higher values represent higher levels of pain (10 = "pain as bad as you can imagine"; 0 = "no pain").
Pain intensity, past week, immediately before intervention session 1. | Immediately before intervention session 1 (study day 1)
  Participants will answer the question "What number best describes your mid and low back pain on average in the past week?". Higher values represent higher levels of pain (10 = "pain as bad as you can imagine"; 0 = "no pain").
Pain intensity, past week, immediately before intervention session 2. | Immediately before intervention session 2 (study day 2, between 48 hours and 2 weeks after study day 1)
  Participants will answer the question "What number best describes your mid and low back pain on average in the past week?". Higher values represent higher levels of pain (10 = "pain as bad as you can imagine"; 0 = "no pain").
Satisfaction with care, immediately after intervention session 1. | Immediately after intervention session 1 (study day 1)
  Participants will answer the question "I am satisfied with the care I received today" with five possible ordinal answers: "Strongly agree", "Agree", "Uncertain", "Disagree", "Strongly disagree" (from The Patient Satisfaction Questionnaire Short-Form [PSQ-18]).
Satisfaction with care, immediately after intervention session 2. | Immediately after intervention session 2 (study day 2, between 48 hours and 2 weeks after study day 1)
  Participants will answer the question "I am satisfied with the care I received today" with five possible ordinal answers: "Strongly agree", "Agree", "Uncertain", "Disagree", "Strongly disagree" (from The Patient Satisfaction Questionnaire Short-Form [PSQ-18]).
Back function - self-reported flexibility, immediately before intervention session 1. | Immediately before intervention session 1 (study day 1)
  Participants will answer the question "How would you rate your back flexibility at the moment?" (adapted from The International Fitness Scale [IFIS]).
Back function - self-reported flexibility, immediately after intervention session 1. | Immediately after intervention session 1 (study day 1)
  Participants will answer the question "How would you rate your back flexibility at the moment?" (adapted from The International Fitness Scale [IFIS]).
Back function - self-reported flexibility, immediately before intervention session 2. | Immediately before intervention session 2 (study day 2, between 48 hours and 2 weeks after study day 1)
  Participants will answer the question "How would you rate your back flexibility at the moment?" (adapted from The International Fitness Scale [IFIS]).
Back function - self-reported flexibility, immediately after intervention session 2. | Immediately after intervention session 2 (study day 2, between 48 hours and 2 weeks after study day 1)
  Participants will answer the question "How would you rate your back flexibility at the moment?" (adapted from The International Fitness Scale [IFIS]).
Back function - self-reported back function, immediately before intervention session 1. | Immediately before intervention session 1 (study day 1)
  Self-reported current back function (numerical rating scale, 0 to 10). Higher values represent higher levels of back function (10 = "Best possible back function", 0 = "Worst possible back function").
Back function - self-reported back function, immediately after intervention session 1. | Immediately after intervention session 1 (study day 1)
  Self-reported current back function (numerical rating scale, 0 to 10). Higher values represent higher levels of back function (10 = "Best possible back function", 0 = "Worst possible back function").
Back function - self-reported back function, immediately before intervention session 2. | Immediately before intervention session 2 (study day 2, between 48 hours and 2 weeks after study day 1)
  Self-reported current back function (numerical rating scale, 0 to 10). Higher values represent higher levels of back function (10 = "Best possible back function", 0 = "Worst possible back function").
Back function - self-reported back function, immediately after intervention session 2. | Immediately after intervention session 2 (study day 2, between 48 hours and 2 weeks after study day 1)
  Self-reported current back function (numerical rating scale, 0 to 10). Higher values represent higher levels of back function (10 = "Best possible back function", 0 = "Worst possible back function").
Back function - self-reported ache, pain, discomfort in the mid and low back, immediately before intervention 1. | Immediately before intervention session 1 (study day 1)
  Ache, pain, discomfort in the mid and low back, by asking "During the past week, have you experienced ache, pain, discomfort in your mid and low back?" (adapted from the Cornell Musculoskeletal Discomfort Questionnaire).
Back function - self-reported ache, pain, discomfort in the mid and low back, immediately before intervention 2. | Immediately before intervention session 2 (study day 2, between 48 hours and 2 weeks after study day 1)
  Ache, pain, discomfort in the mid and low back, by asking "During the past week, have you experienced ache, pain, discomfort in your mid and low back?" (adapted from the Cornell Musculoskeletal Discomfort Questionnaire).
Participant's reasons for beliefs about intervention assigned, immediately after intervention session 1. | Immediately after intervention session 1 (study day 1)
  Following the blinding assessment for the primary and secondary outcomes, participants will be asked the free text question, "Why do you believe you received this treatment?".
Participant's reasons for beliefs about intervention assigned, immediately after intervention session 2. | Immediately after intervention session 2 (study day 2, between 48 hours and 2 weeks after study day 1)
  Following the blinding assessment for the primary and secondary outcomes, participants will be asked the free text question, "Why do you believe you received this treatment?".
Outcome assessor's reasons for beliefs about intervention assigned, immediately after intervention session 1. | Immediately after intervention session 1 (study day 1)
  Following the blinding assessment for the primary and secondary outcomes, outcome assessors will be asked the free text question, "Why do you believe this participant received this treatment?".
Outcome assessor's reasons for beliefs about intervention assigned, immediately after intervention session 2. | Immediately after intervention session 2 (study day 2, between 48 hours and 2 weeks after study day 1)
  Following the blinding assessment for the primary and secondary outcomes, outcome assessors will be asked the free text question, "Why do you believe this participant received this treatment?".
Participant credibility/expectancy of active and control interventions, as measured with the credibility/expectancy questionnaire, immediately after intervention session 2. | Immediately after intervention session 2 (study day 2, between 48 hours and 2 weeks after study day 1)
  Participants will complete the six items from the credibility/expectancy questionnaire with a hypothetical scenario: "For the following six questions, imagine that you were experiencing uncomfortable low back pain and were exposed to the treatment you received for a period of about 8 weeks." Item 1: "At this point, how logical would the SMT treatment offered to you seem?" Item 2: "At this point, how successful do you think this SMT treatment would be in reducing your symptoms?" Item 3: "How confident would you be in recommending this SMT treatment to a friend experiencing similar symptoms?" Item 4: "By the end of the SMT treatment period, how much improvement in your symptoms do you think would occur?" Item 5: "At this point, how much do you really feel that this SMT treatment would help you to reduce your symptoms?" Item 6: "By the end of the SMT period, how much improvement in your symptoms do you really feel would occur?" Higher values represent higher credibility and expectancy.

CONTACTS AND LOCATIONS:
Overall Officials: Cesar A Hincapié, DC PhD, Principal Investigator — Balgrist University Hospital and University of Zurich
Locations (1):
- Balgrist University Hospital and CHIROMED Praxis im Seefeld, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
The central contact person and principal investigator will make supporting information available upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code

REFERENCES:
- [Derived] Munoz Laguna J, Kurmann A, Hofstetter L, Nyantakyi E, Braun J, Clack L, Bang H, Farshad M, Foster NE, Puhan MA, Hincapie CA; SALuBRITY Blinding Clinician Group. 'Which treatment do you believe you received?' A randomised blinding feasibility trial of spinal manual therapy. Chiropr Man Therap. 2025 Jan 14;33(1):4. doi: 10.1186/s12998-024-00561-0. PMID 39810207
- [Derived] Munoz Laguna J, Kurmann A, Hofstetter L, Nyantakyi E, Clack L, Bang H, Foster NE, Braun J, Puhan MA, Farshad M, Hincapie CA. Feasibility of blinding spinal manual therapy interventions among participants and outcome assessors: protocol for a blinding feasibility trial. Pilot Feasibility Stud. 2024 May 2;10(1):70. doi: 10.1186/s40814-024-01492-6. PMID 38698433